CLINICAL TRIAL: NCT03206645
Title: Phase 1B Trial With Unesbulin in High-Grade Serous Ovarian Cancer: a Targeted Approach Toward Chemoresistant Stem-Like Cancer Cells
Brief Title: Unesbulin in Women With Ovarian Cancer Receiving Neoadjuvant Chemotherapy
Acronym: PTC-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-PTC-001
Record Dates: First submitted 2017-06-01; First posted 2017-07-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — PTC596

STUDY DESIGN:
Intervention Model Description: This trial will utilize a traditional 3+ 3 design with dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin/Paclitaxel + PTC596 (Experimental): Carboplatin AUC 6mg/L IV on day 1; Paclitaxel 175mg/m2 IV on day 1; Unesbulin PO, twice a week, on day 1, 4, 8, 11, 15 and 18 per 21-day cycle for the first 3 cycles.
  Interventions: Drug: Unesbulin

INTERVENTIONS:
Drug: Unesbulin — Unesbulin will be given in combination with carboplatin and paclitaxel for up to 7 cycles depending on which cohort the patient is in.
  Other Names: PTC596

SUMMARY:
This is an open-label Phase Ib dose-escalation study to determine the safety, tolerability, and pharmacokinetics of Unesbulin when combined with and following conventional chemotherapy and as maintenance therapy as a capsule (weight based dosing) and a tablet (fixed dosing) in women with epithelial ovarian, fallopian tube or primary peritoneal cancer which is previously untreated.

DETAILED DESCRIPTION:
For all cohorts, the study drug Unesbulin will be orally administered prior to chemotherapy (paclitaxel and carboplatin), twice a week of each 21-day cycle. Chemotherapy will be administered on day 1 of each cycle by vein. Dose escalation levels for Unesbulin will occur per protocol and doses may be de-escalated for management of toxicity. Patients will receive a total of 3 cycles of Unesbulin and chemotherapy. Surgery will be performed within 6 weeks after the last dose of Cycle 3. An additional 3-7 cycles of Unesbulin and chemotherapy (carboplatin and paclitaxel) may be given as maintenance therapy for up to two years at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented epithelial ovarian, primary peritoneal or fallopian tube carcinoma or high grade serous adenocarcinoma, endometrioid adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma,or adenocarcinoma not otherwise specified (N.O.S.)
* Newly diagnosed and be previously untreated
* Adequate bone marrow function, renal function, and hepatic function
* Baseline neuropathy (sensory and motor) less than or equal to Grade 1
* Free of active infection requiring parenteral antibiotics or a serious uncontrolled medical illness or disorder within four weeks of study entry.
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration. Continuation of hormone replacement therapy is permitted.
* Have a performance status score of 0, 1, or 2 by Eastern Cooperative Group (ECOG) criteria.
* Patients of childbearing potential must have a negative pregnancy test prior to the study entry and be practicing an effective form of contraception. If applicable, patients must discontinue breastfeeding prior to study entry.

Exclusion Criteria:

* Prior treatment with Unesbulin or standard of care drugs (cis- or carboplatin or paclitaxel.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Unesbulin or other agents used in this study.
* Have a clinical requirement for ongoing systemic immunosuppressive therapy such as chronic steroid use not related to chemotherapy administration.
* Receiving treatment for active autoimmune disease including systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease and rheumatoid arthritis.
* History of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies within the last three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy. Patients with concomitant endometrial cancer diagnosed at the time of their ovarian cancer are allowed to participate if the endometrial cancer is FIGO stage IB or less.
* Prior radiotherapy to any portion of the abdominal cavity or pelvis. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted if completed more than three years prior to registration and the patient remains free of recurrent or metastatic disease.
* Prior chemotherapy for any abdominal or pelvic tumor. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* Known active hepatitis, ongoing systemic bacterial, fungal, or viral infection; known human immunodeficiency virus (HIV) infection or acquired-immunodeficiency syndrome (AIDS)-related illness.
* Have concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or expose the patient to extreme risk or decreased life expectancy.
* Have childbearing potential but not practicing adequate contraception, or pregnant, or breastfeeding.
* History or active CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months prior to study treatment.
* Concomitant therapy with any of the following: other non-study cytotoxic chemotherapy; other investigational therapies.
* Prior bone marrow/hematopoietic stem cell transplantation
* Use of an investigational drug within 4 weeks of dosing in the current study
* History of major surgical procedure within 28 days prior to start of study treatment
* Presence of history of moderate to severe pulmonary dysfunction (e.g., moderate/severe chronic obstructive pulmonary disease, post-pneumoectomy, shortness of breath with limited exertion).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and dose limiting toxicities | 42 days
  To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of Unesbulin in combination with and following conventional chemotherapy and as maintenance as a capsule (weight-based dosing) and a tablet (fixed dosing). Standard chemotherapy will be comprised of carboplatin and weekly paclitaxel. The DLTs will be based on adverse events that occur during administration of the first 2 cycles of combination Unesbulin and chemotherapy (a cycle = 21 days).
Number of patients able to tolerate drug combination | 3 years
  To examine the tolerability of the combination at the MTD of Unesbulinassessed in combination with standard neoadjuvant chemotherapy.
Phase 2 Dose | 3 years
  To determine the recommended phase II dose (RP2D) of Unesbulin in combination with standard neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Evaluate clinical response | 3 years
  Evaluate clinical response by measuring serum CA-125. If CA-125 is initially above the upper normal limit, it must normalize for patients to be considered in complete clinical response.
Evaluate pharmacokinetic Area Under the Curve (AUC) | 3 months
  To evaluate pharmacokinetic parameters of Unesbulin in patients with stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer receiving neoadjuvant chemotherapy with carboplatin/paclitaxel
Evaluate pharmacokinetic Maximum Concentration observed (Cmax) | 3 months
  To evaluate pharmacokinetic parameters of Unesbulin in patients with stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer receiving neoadjuvant chemotherapy with carboplatin/paclitaxel
Evaluate pharmacokinetic Time of Maximum Concentration observed (Tmax) | 3 months
  To evaluate pharmacokinetic parameters of Unesbulin in patients with stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer receiving neoadjuvant chemotherapy with carboplatin/paclitaxel
Evaluate pharmacokinetic half life (t1/2) | 3 months
  To evaluate pharmacokinetic parameters of Unesbulin in patients with stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer receiving neoadjuvant chemotherapy with carboplatin/paclitaxel
Progression free survival | one year
  The duration of time (one year) that patients are alive and their cancer is progression-free.
Progression free survival | two years
  The duration of time (two years) that patients are alive and their cancer is progression-free.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Study Chair — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No